CLINICAL TRIAL: NCT04298541
Title: SSTR2-Targeted PET Imaging of Meningioma: Direct Comparison of Ga-68-DOTATATE and Ga-68-DOTATOC
Brief Title: Direct Comparison of Ga-68-DOTATATE and Ga-68-DOTATOC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-10021002
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Intervention Model Description: The study intervention consists of 2 PET scans that will be performed at least 24h apart using 68-Ga-DOTATATE and 68-Ga-DOTATOC radiotracers, in patients with suspected meningioma that are planned for subsequent surgery.
  Visit 1 Patients will undergo a 68-Ga-DOTATATE PET/CT or PET/MR scan as standard of care, or as part of a separate research study.
  Visit 2 At least 24h and up to 4 weeks apart from Visit 1, patients will undergo 68Ga-DOTATOC PET/CT scan.
  Follow-up Phase Patients enrolled in the study are planned for surgery as part of SOC. After the two scans, patients will undergo surgery and a histopathologic analysis of the resected tumor will be performed. The histopathology results will be used to correlate molecular biomarkers with imaging parameters. During the follow up period a review of clinical and imaging records related to the diagnosis will be conducted by the research team as part of the study during the follow- up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Meningioma (Experimental): Subjects with suspected meningioma planned for surgery who meet the inclusion and exclusion criteria.
  Interventions: Drug: Ga-68- DOTATATE; Drug: Ga-68-DOTATOC

INTERVENTIONS:
Drug: Ga-68- DOTATATE — The study intervention consists of two PET scans that will be performed using two different radiotracers, 68-Ga-DOTATATE and 68-Ga-DOTATOC. Ga-68-DOTATATE and 68-Ga-DOTATOC are PET radiotracers targeting somatostatin receptors.
  The study intervention consists of 2 PET scans that will be performed at least 24h apart using 68-Ga-DOTATATE and 68-Ga-DOTATOC radiotracers, in patients with suspected meningioma that are planned for subsequent surgery.
Drug: Ga-68-DOTATOC — The study intervention consists of two PET scans that will be performed using two different radiotracers, 68-Ga-DOTATATE and 68-Ga-DOTATOC. Ga-68-DOTATATE and 68-Ga-DOTATOC are PET radiotracers targeting somatostatin receptors.
  The study intervention consists of 2 PET scans that will be performed at least 24h apart using 68-Ga-DOTATATE and 68-Ga-DOTATOC radiotracers, in patients with suspected meningioma that are planned for subsequent surgery.

SUMMARY:
The goal of this study is to propose the first direct comparison of Ga-68-DOTATATE PET/CT or PET/MR and Ga-68-DOTATOC PET/CT in patients with meningioma.

DETAILED DESCRIPTION:
The investigator is proposing a direct comparison of Ga-68-DOTATATE and -DOTATOC in a pilot cohort of patients with meningioma, and hypothesize non-inferiority of DOTATOC. This pilot study will form the basis for a subsequent prospective clinical trial and will allow us to optimize our existing imaging protocols, while developing a more cost-effective protocol.

Primary Objectives:

* Optimize the Ga-68-DOTATOC PET/CT protocol.
* Compare Ga-68-DOTATATE PET and -DOTATOC PET/CT in patients with meningioma.

Secondary Objectives

• Correlate Ga-68-DOTATATE PET and -DOTATOC PET/CT with clinical and pathological characteristics

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with clinically suspected meningioma
* Patients planned for surgery - undergoing preoperative workup
* No contraindications to either radiotracer

Exclusion Criteria:

* Age less than 18 years
* Inability to lay on the scanner table for the required period of time, e.g., due to bone pain or claustrophobia.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Qualitatively measure the visual appearance of target lesion to cranial blood pool using the maximum SUV ratio to compare results from Ga-68-DOTATATE and -DOTATOC PET. | Over 12 months
  Compare visual appearance qualitatively using the maximum SUV ratio of target lesion to cranial blood pool (i.e. superior sagittal sinus reference region) of DOTATATE and DOTATOC PET scans in patients with meningioma.
  Based on our pilot clinical case series, the following reference regions will be evaluated:
  1. Suspected meningioma;
  2. Pituitary gland;
  3. Superior sagittal sinus;
  4. Brain parenchyma.
  Dynamic PET will be acquired and data will be analyzed including comparison of tissue-activity curves and Patlak analysis, as established by the PI in a pilot cohort.
  Extent of meningioma based on Ga-68-DOTATATE- and DOTATOC PET/CT will be compared to extent of disease as determined by MRI.
Quantitatively measure the visual appearance of target lesion to cranial blood pool using the maximum SUV ratio to compare results from Ga-68-DOTATATE and -DOTATOC PET. | Over 12 months
  Compare visual appearance quantitatively using the maximum SUV ratio of target lesion to cranial blood pool (i.e. superior sagittal sinus reference region) of DOTATATE and DOTATOC PET scans in patients with meningioma.
  Qualitative analysis will include evaluation by board certified radiologists with expertise in nuclear medicine/ molecular imaging who will be blinded to the radiotracer injected. Quantitative analysis will include extraction of the ratio of lesion's SUVmax values/reference regions.

SECONDARY OUTCOMES:
Compare molecular biomarker (Ki67) analysis to Ga-68-DOTATATE PET and Ga-68-DOTATOC PET by measuring biomarker histopathology (Ki67) results to the maximum SUV ratio of target lesion to cranial blood pool. | Over 12 months
  Patients enrolled in the study will subsequently undergo surgical resection of the lesion. The surgical specimen will be used for biomarker analysis to assess genetic information. The additional staining that will take place for research purposes includes, specifically Ki67. These parameters will be correlated with parameters acquired from the 68-Ga-DOTATATE and - DOTATOC PET scans.
Compare molecular biomarker (EGFR) analysis to Ga-68-DOTATATE PET and Ga-68-DOTATOC PET by measuring biomarker histopathology (EGFR) results to the maximum SUV ratio of target lesion to cranial blood pool. | Over 12 months
  Patients enrolled in the study will subsequently undergo surgical resection of the lesion. The surgical specimen will be used for biomarker analysis to assess genetic information. The additional staining that will take place for research purposes includes, specifically (epidermal growth factor receptor, EGFR). These parameters will be correlated with parameters acquired from the 68-Ga-DOTATATE and - DOTATOC PET scans.
Compare molecular biomarker (progesterone receptor) analysis to Ga-68-DOTATATE PET and Ga-68-DOTATOC PET by measuring biomarker histopathology (progesterone receptor) results to the maximum SUV ratio of target lesion to cranial blood pool. | Over 12 months
  Patients enrolled in the study will subsequently undergo surgical resection of the lesion. The surgical specimen will be used for biomarker analysis to assess genetic information. The additional staining that will take place for research purposes includes, specifically progesterone receptor. These parameters will be correlated with parameters acquired from the 68-Ga-DOTATATE and - DOTATOC PET scans.
Compare molecular biomarker (SSTR2 expression) analysis to Ga-68-DOTATATE PET and Ga-68-DOTATOC PET by measuring biomarker histopathology (SSTR2 expression) results to the maximum SUV ratio of target lesion to cranial blood pool. | Over 12 months
  Patients enrolled in the study will subsequently undergo surgical resection of the lesion. The surgical specimen will be used for biomarker analysis to assess genetic information. The additional staining that will take place for research purposes includes, specifically SSTR2 expression. These parameters will be correlated with parameters acquired from the 68-Ga-DOTATATE and - DOTATOC PET scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Ivanidze, MD/Ph.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No